CLINICAL TRIAL: NCT02765620
Title: PERCIST Criteria for Response Evaluation of Non-surgical Therapy in Patients With Solid Tumors:Prospective Multicenter Study
Brief Title: PERCIST Criteria for Response Evaluation With Solid Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Shengjing Hospital (Other); First Affiliated Hospital of Jinan University (Other); Harbin Medical University (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: ED12345
Record Dates: First submitted 2016-04-11; First posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-03

CONDITIONS: Lung Neoplasms; Breast Neoplasms; Colonic Neoplasms; Lymphoma
Keywords: Positron-Emission Tomography; Response Criteria; solid tumor
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Colonic Neoplasms; Lymphoma | interventions — Radiation-Protective Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- drug: Early treatment response assessment: using baseline data and early follow-up data Evaluate treatment response: using baseline data, early follow-up data and final data Compare PERCIST to RECIST criteria: correlation analysis Evaluate prognostic value: using baseline data, early follow-up data, final data as well as follow up PFS and OS time (Kaplan-Meier survival plot
  Interventions: Other: drug&radiation
- radiation: Early treatment response assessment: using baseline data and early follow-up data Evaluate treatment response: using baseline data, early follow-up data and final data Compare PERCIST to RECIST criteria: correlation analysis Evaluate prognostic value: using baseline data, early follow-up data, final data as well as follow up PFS and OS time (Kaplan-Meier survival plot
  Interventions: Other: drug&radiation

INTERVENTIONS:
Other: drug&radiation — 1. Early treatment response assessment: using baseline data and early follow-up data
  2. Evaluate treatment response: using baseline data, early follow-up data and final data
  3. Compare PERCIST to RECIST criteria: correlation analysis
  4. Evaluate prognostic value: using baseline data, early follow-up data, final data as well as follow up PFS and OS time (Kaplan-Meier survival plot)

SUMMARY:
Chemo-radiotherapy and targeted therapy are widely used as non-surgical treatments for solid tumors. Early assessment of treatment response is considered efficient and helpful to clinical management and personalized therapy.RECIST 1.1 criteria was accepted widely. Complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD) are defined in the RECIST criteria. This type of classification divides intrinsically continuous data (tumor size) into 4 bins, losing statistical power for ease of nomenclature and convenience. The 18F-FDG PET exam is based on metabolic information and considered to overcome limitations of anatomic imaging and more suitable for assessment of therapeutic response.PERCIST 1.0 proposes a series of detailed and unambiguous regulations about standardization procedures to ensure the reproducibility. Complete metabolic response (CMR), partial metabolic response (PMR), stable metabolic disease (SMD), and progressive metabolic disease (PMD) are defined in the PERCIST criteria.

So far, there have several studies using metabolic-based PERCIST criteria in patients with solid tumors, including lung cancer, digestive tumor and lymphoma, etc. But all of these studies had limitations of small study sample, thus were need to be further investigated. Compared to RECIST, the advantages of PERCIST were to evaluate chemotherapy, especially targeted therapy, to distinguish PMR and SMD patients from SD group in RECIST, and to better predict the response rate. Recently, several studies applied PERCIST criteria to evaluate neoadjuvant chemotherapy in pancreatic cancer and rectal cancer, and revealed the metabolic response results were well related to pathology. All these studies conclude PERCIST criteria could help making clinical therapeutic decisions. Moreover, several studies have shown that PERCIST has advantage in predicting early response of several malignant tumors.

The aim of this multicenter study is 1) to evaluate treatment response in newly diagnosed and pre-therapeutic patients with solid tumors who are going to receive a baseline , an early follow-up (after a certain period of treatment cycle) and a final (after treatment) 18F-FDG PET/CT; 2) to compared PERCIST criteria to RECIST 1.1 criteria in prediction treatment response, especially in early stage of treatment; 3) to reveal the value of PERCIST criteria in clinical therapeutic management and tailed therapy.

DETAILED DESCRIPTION:
1. Newly diagnosed and pre-therapeutic patients with solid tumors, including but not limited to: lung cancer, lymphoma, gastric cancer, breast cancer, colorectal cancer, ovarian cancer, cervical cancer etc.
2. Study sample: based on ongoing retrospective results, the optimal study sample is expected to be >150 cases per each cancer type.
3. Treatment regimen: based on certain cancer type.
4. Inclusion criteria: age 30-80 years old ( might differ based on certain cancer type) ; newly diagnosis of solid tumor proved by imaging; pathology proved to be primary solid tumor; first PET/CT scan was performed before any kinds of anti-tumor treatment including surgery; no other anti-tumor treatments except for that required during the trial; written and informed consent with signature before the study; complete medical history and clinical record (including physical examination, electrocardiogram, hematology, biochemistry, tumor pathology etc); follow-up of PSF and OS over a year
5. Exclusion criteria: pregnancy, lactation, and impaired renal or liver function; receive additional anti-tumor treatments (including surgery) other than that required during the trial; poorly controlled diabetes; poor compliance; failed to perform scans; contrary to the standard operating procedures; without a definite pathologic diagnosis or follow-up results; not suitable for clinical trials (for example with mental illness)
6. Withdrawal criteria: subjects demand; miss follow-ups; severe incident; other reasons that failed to complete the trial

Prospective Study:

18F-FDG PET/CT scans were performed before treatment (baseline), after a certain period of treatment cycle (early follow-up) and after the whole treatment process (final). Using PERCIST 1.0 criteria in PET imaging and RECIST 1.1 criteria in CT imaging to monitor and assess treatment response and prognosis.

1. Early treatment response assessment: using baseline data and early follow-up data Base on PERCIST 1.0 criteria, CMR, PMR and SMD were considered response; PMD was considered non-response; Base on RECIST 1.1 criteria, CR, PR, SD were considered response; PD considered non-response
2. Evaluate treatment response: using baseline data, early follow-up data and final data Base on PERCIST 1.0 criteria, CMR, PMR and SMD were considered response; PMD was considered non-response; Base on RECIST 1.1 criteria, CR, PR, SD were considered response; PD considered non-response
3. Compare PERCIST to RECIST criteria: correlation analysis
4. Evaluate prognostic value: using baseline data, early follow-up data, final data as well as follow up PFS and OS time (Kaplan-Meier survival plot)

Study protocol

1)Clinical data: enroll patients according to inclusion/exclusion criteria, record all clinical information and imaging data and keep to follow-up over one year.

2)18F-FDG PET/CT protocol: GE Discovery Elite PET/CT scanner was used in multicenter trials with the same protocol. Patients were instructed to fast for at least 6 hours before 18F-FDG PET/CT scan. Blood glucose level was measured before tracer was injected. Whole-body PET/CT images, generally from the top of the skull to mid-thigh, were acquired 50~70 min after intravenous injection of 18F-FDG at the dose of 0.08~0.10 mCi per kilograms of body weight. Patients were asked to void their bladder immediately before scanning to minimize the presence of the tracer in the urinary tract. PET data were acquired and reconstructed using SharpIR+ VUE Point HD+TOF, 2min/bed. The PET data were attenuation corrected (AC) by the integrated CTAC technology. CT data were acquired in breath-hold with 120 kV, 30-210 mA modulated by GE SmartmA technique with a noise index of 25; with slice thickness 3.75 mm, slice interval 3.27 mm, pitch 1.375, matrix size 512×512 and scan FOV 50cm.

3)Data archive: All clinical information and original DICOM data were archived in individual institution. Post-processed results using PETVCAR software were archived and uploaded to central server. Institutions without PETVCAR software need to uploaded PET/CT DICOM data to central server which will be analysis by a certain physician.

4)Data Analysis: patient imaging data were analysis by more than three professional nuclear medicine physicians in GE Advantage Workstation (AW) using PETVCAR software (based on RECIST 1.1 criteria and PERCIST 1.0 criteria).

Fig 1. RECIST1.1 and PERCIST1.0 criteria in PETVCAR software

RECIST 1.1 criteria:

Measurable, unidimensional (LD only: size with conventional techniques≥20 mm, with spiral CT≥10 mm; nodes: target short axis ±15 mm, nontarget 10- to 15-mm nodes, normal< 10 mm)

Nonmeasurable: all other lesions, including small lesions; evaluable is not recommended

Target lesions (change in sum of LDs, maximum of 2 per organ up to 5 total [more than 1 organ]):

CR, disappearance of all target lesions, confirmed at ≥4 wk; PR, ≥30% decrease from baseline, confirmed at 4 wk; PD, ≥20% increase over smallest sum observed and overall 5-mm net increase or appearance of new lesions; SD, neither PR nor PD criteria met

Nontarget lesions:

CR, disappearance of all nontarget lesions and normalization of tumor markers, confirmed at ≥4 wk; PD, unequivocal progression of nontarget lesions or appearance of new lesions; non-PD: persistence of one or more nontarget lesions or tumor markers above normal limits; PD must be ''unequivocal'' in nontarget lesions (e.g., 75% increase in volume); PD can also be new ''positive PET'' scan with confirmed anatomic progression. Stably positive PET is not PD if it corresponds to anatomic non-PD

PERCIST 1.0 criteria:

For target lesions:

CMR: complete resolution of 18F-FDG uptake within measurable target lesion so that it is less than mean liver activity and indistinguishable from surrounding background blood-pool levels. Disappearance of all other lesions to background bloodpool levels. Percentage decline in SUL should be recorded from measurable region, as well as (ideally) time in weeks after treatment was begun. No new 18F-FDG-avid lesions in pattern typical of cancer. If progression by RECIST, must verify with follow-up.

PMR: reduction of minimum of 30% in target measurable tumor 18F-FDG SUL peak. Absolute drop in SUL must be at least 0.8 SUL units, as well. Measurement is commonly in same lesion as baseline but can be another lesion if that lesion was previously present and is the most active lesion after treatment. ROI does not have to be in precisely same area as baseline scan, though typically it is. No increase, .30% in SUL or size of target or nontarget lesions (i.e., no PD by RECIST or IWC) (if PD anatomically, must verify with follow-up). Reduction in extent of tumor 18F-FDG uptake is not requirement for PMR. Percentage decline in SUL should be recorded, as well as (ideally) time in weeks after treatment was begun (i.e., PMR 240, 3). No new lesions.

SMD: not CMR, PMR, or PMD. SUL peak in metabolic target lesion should be recorded, as well as (ideally) time from start of most recent therapy, in weeks (i.e., SMD 215, 7).

PMD: 30% increase in 18F-FDG SUL peak, with .0.8 SUL unit increase in tumor SUV peak from baseline scan in pattern typical of tumor and not of infection/treatment effect. OR: Visible increase in extent of 18F-FDG tumor uptake (75% in TLG volume with no decline in SUL. OR: New 18F-FDG-avid lesions that are typical of cancer and not related to treatment effect or infection. PMD other than new visceral lesions should be confirmed on follow-up study within 1 mo unless PMD also is clearly associated with progressive disease by RECIST 1.1. PMD should be reported to include percentage change in SUV peak, (ideally, time after treatment, in weeks) and whether new lesions are present/absent and their number (i.e., PMD, 135, 4, new: 5). Because SUL is continuous variable, dividing response criteria into limited number of somewhat arbitrary response categories loses much data. For this reason, PERCIST preserves percentage declines in SUV peak in each reported category. Because rapidity with which scan normalizes is important (faster appears better), PERCIST asks for time from start of treatment as part of reporting. For example, CMR 90, 1, is probably superior to CMR 90, 10, especially if latter patient were SMD 20, 1. More than one measurement of PET response may be needed at differing times, and it may be treatment type-dependent. PERCIST 1.0 evaluates SUL peak of only hottest tumor. This is possible limitation of approach, but lesions and their responses are highly correlated in general. Additional data are required to determine how many lesions should be assessed over 1. A suggested option is to include the 5 hottest lesions, or the 5 observed on RECIST 1.1 that are most measurable. Percentage change in SUL can be reported for single lesion with largest increase in uptake or smallest decline in uptake. Additional studies will be needed to define how many lesions are optimal for assessment.

For nontarget lesions:

CMR, disappearance of all 18F-FDG-avid lesions: PMD, unequivocal progression of 18F-FDG-avid nontarget lesions or appearance of new 18F-FDG-avid lesions typical of cancer; non-PMD: persistence of one or more nontarget lesions or tumor markers above normal limits.

5)Follow-ups: including clinical changes (weight, pain) before and after treatment, treatment regimen, biochemistry result, pathological result, immunohistochemical result; PFS and OS time

Quality control:

1. All PET/CT scans were performed in GE Discovery Elite scanner.
2. Reproducibility and accuracy of each institution were analysis by third party using a PET NEMA phantom.
3. Multiple PET/CT scans of one patient were controlled by Q-Check software to make sure the data quality for PETVCAR analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80 years old ( might differ based on certain cancer type)
* Newly diagnosis of solid tumor proved by imaging
* Pathology proved to be primary solid tumor
* First PET/CT scan was performed before any kinds of anti-tumor treatment including surgery
* No other anti-tumor treatments except for that required during the trial
* Written and informed consent with signature before the study
* Complete medical history and clinical record (including physical examination, electrocardiogram, hematology, biochemistry, tumor pathology etc)
* Follow-up of PSF and OS over a year

Exclusion Criteria:

* Pregnancy, lactation, and impaired renal or liver function
* Receive additional anti-tumor treatments (including surgery) other than that required during the trial
* Poorly controlled diabetes
* Poor compliance
* Failed to perform scans
* Contrary to the standard operating procedures
* Without a definite pathologic diagnosis or follow-up results
* Not suitable for clinical trials (for example with mental illness)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed and pre-therapeutic patients with solid tumors, including but not limited to: lung cancer, lymphoma, gastric cancer, breast cancer, colorectal cancer, ovarian cancer, cervical cancer etc.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-01 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate treatment response by PERCIST to RECIST 1.1 criteria in early stage of treatment | about 4 weeks
  Cycle 2 (each cycle is 10 days)
Evaluate treatment response by PERCIST to RECIST 1.1 criteria after the whole treatment process | about 6 months

SECONDARY OUTCOMES:
PFS | up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes